CLINICAL TRIAL: NCT04163302
Title: Safety and Efficiency Study of CD19-PD1-CART Cell in Relapsed/Refractory B Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Quanshun Wang, Chief of Hematology Department of Hainan Hospital of PLA General Hospital; Vice Chief of Hematology Department of PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNYY-XYK-02
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma, B-Cell
Keywords: Lymphoma; Chimeric antigen receptor T cell; Chimeric antigen receptor; Immunotherapy; PD-1; CD19
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Intervention Model Description: This study was a single-center, open-label, single-arm, non-randomized clinical trial, which was divided in 3 groups by different infusion dose level. Firstly, each dose group has 3 patients. The pretreatment regimen of cyclophosphamide (25mg/m2 for 3 consecutive days) and fludarabine (10mg/kg for 3 consecutive days) was given before CART cells were reinfused. CART cells were reinfused on the third day after the pretreatment. If no serious side effects emerges in the group, then the next group uses the subsequent higher dose. If serious side effects emerges in a single patients in any dose level, 3 more patients will be enrolled to the same dose level. After 9 or more patients, the investigators select the safest dose and recruit more patients for CART test to explore its effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19+ Lymphoma (Experimental): This study is to evaluate the efficacy and safety of CD19-PD1-CART cells therapy for patients with Relapsed/Refractory B Cell Lymphoma.
  Interventions: Biological: CD19-PD1-CART Cell

INTERVENTIONS:
Biological: CD19-PD1-CART Cell — This study was a single-center, open-label, single-arm, non-randomized clinical trial, which has 3 groups by infusion dose level. Firstly, each dose group has 3 patients. The pretreatment regimen of cyclophosphamide (25mg/m2 for 3 consecutive days) and fludarabine (10mg/kg for 3 consecutive days) was given before CART cells were reinfused. CART cells were reinfused on the third day after the pretreatment. If no serious side effects emerges in the group, then the next group uses the subsequent higher dose. If serious side effects emerges in a single patients in any dose level, 3 more patients will be enrolled to the same dose level. After 9 or more patients, the investigators select the safest dose and recruit more patients for CART test to explore its effectiveness.

SUMMARY:
This is a single center, non-randomized, open-label, phase 2 study to evaluate the efficacy and safety of CD19-PD1-CART cells therapy for patients with relapsed/refractory B Cell Lymphoma.

DETAILED DESCRIPTION:
Lymphoma is a malignant tumor originating from lymph nodes or other lymphoid tissues. It can be divided into B cells, T cells, and NK cell lymphomas depending on the origin of different lymphocytes. Among them, B cell lymphoma accounts for about 90% of lymphoma.

Chimeric antigen receptor T (CART) cells is a promising treatment for lymphoma. T lymphocytes from patients are separated and engineered with CD19-CAR, to specifically recognize and eliminate CD19-positive tumor cells. At present, many CD19CART cells therapy studies are in the stage of clinical research and have achieved significant clinical effects.

Although there are some CD9CART cells clinical trials, the therapeutic effect on lymphoma is significantly lower than that of acute leukemia. One of the reasons is that lymphoma has the nature of solid tumors, whichi has a certain immunosuppressive microenvironment. The clinical trials of anti-PD-1 antibody drugs against lymphoma also show good therapeutic efficacy. Therefore, the combination of anti-PD-1 or PD-L1 antibody and CD19CART is one of the ways to improve the therapeutic effect of CART cells.

The investigators screened PD-1 mutants that have high bind with the PD-L1 ligand, and prepared CD19CART which secretes the mutant PD-1Fc fusion protein. Preclinical studies have shown that CD19CART cells secreting mutant PD-1Fc fusion protein have a superior killing effect to CD19CART cells which does not express PD-1 fusion protein.

The trial was conducted to explore the safety and efficacy of CD19-PD1-CART cells in Relapsed/Refractory B Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 14 to 80 years (including 14 and 80 years old).
2. The diagnosis was Refractory/relapsed B-cell lymphoma.(Meeting 1 of the first 4 items plus item 5)

   A.Tumor shrinkage less than 50% or disease progression after 4 cycles of standard chemotherapy.

   B.Achieved CR after standard chemotherapy, but relapsed within 6 months.

   C.2 or more relapses after CR.

   D.Not suitable for HSCT, or relapse after HSCT.

   E.Subjects must have received adequate treatment in the past and the predicted survival is more than three months.
3. Patient or his or her legal guardian voluntarily participates in this stuy and signs an informed consent form.
4. Flow cytometry or immunohistochemistry showed CD19 positive in tumor cells.
5. No serious concomitant disease and major organ function is not serious abnormal.
6. ECOG physical condition score 0-3 or KPS score > 80.
7. the test meets the following indicators:

A.ALT/AST < 2.5 times the upper limit of normal (ULN) and total bilirubin≤34.2μmol/L.

B.Creatinine < 176.8 μmol/L.

C.WBC≥2.5×109/L ，LY≥0.7×109/L，LY%≥15%.

D.PT/INR < 1.7 or PT was extended by less than 4 seconds.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Patients whose tumor cell don't have positive CD19 antigen.
3. Active hepatitis B or hepatitis C, HIV/AIDS infection, any uncontrolled active infection.
4. Patients who are using steroid drugs throughout the body currently.
5. Patients who have received any gene therapy in the past.
6. Patients who are allergy to immunotherapy and related drugs.
7. Patients with heavy heart disease or poorly controlled high blood pressure.
8. Patients who received chemotherapy or radiation 4 weeks before the study began.
9. Patients who are participating in other clinical trials.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 3 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Overall Remission Rate(ORR) of CD19-PD1-CART cells in Lymphoma | 3 years
  ORR will be assessed from the first CAR-T cell infusion to death or last follow-up
Overall survival(OS) of CD19-PD1-CART cells in Lymphoma | 3 years
  OS will be assessed from the first CAR-T cell infusion to death or last follow-up
Progress-free survival(PFS) of CD19-PD1-CART cells in Lymphoma | 3 years
  PFS will be assessed from the first CAR-T cell infusion to death or last follow-up
Rate of CD19-PD1-CARTcells in peripheral blood cells | 3 years
  In vivo (peripheral blood) rate of CD19-PD1-CART cells were determined by means of flow cytometry.
Quantity of CD19-PD1-CART cells copies in peripheral blood cells. | 3 years
  In vivo (peripheral blood) quantity of CD19-PD1-CART cells copies copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Quanshun Wang, Study Chair — Hainan Hospital of Chinese PLA General Hospital; Wengshuai Zheng, Study Director — Hainan Hospital of Chinese PLA General Hospital; Lixun Guan, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Lu Wang, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Yuanyuan Xu, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Yalei Hu, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital; Zhengyang Gu, Principal Investigator — Hainan Hospital of Chinese PLA General Hospital
Locations (1):
- Hai Nan Hospital of Chinese PLA General Hospital, Sanya, Hainan, China

IPD SHARING:
Plan to Share IPD: No